CLINICAL TRIAL: NCT05672472
Title: Clinical Study of Neutrophil Elastase Inhibitor in Treatment of Acute Respiratory Distress Syndrome Patients With Mechanical Ventilation Caused by Sepsis
Brief Title: Neutrophil Elastase Inhibitor in Treatment of ARDS Patients With Mechanical Ventilation Caused by Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yuting Li, Attending doctor, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yuting Li1
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome; Sepsis; Neutrophil elastase inhibitor; Mechanical ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Sepsis | interventions — Respiration, Artificial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sivelestat sodium (Experimental): The patients in the test group were given 0.2 mg/kg. h of sivelestat sodium (0.1 g/tube, Shanghai Huilun Jiangsu Pharmaceutical Co., Ltd.) (the daily dose was added to 250 ml of 0.9% sodium chloride) intravenously for 24 hours and 5 consecutive days.
  Interventions: Drug: Sivelestat sodium
- sodium chloride (Placebo Comparator): The patients in the control group were given 250 ml 0.9% sodium chloride (250ml/bag, Jilin Dubang Pharmaceutical Co., Ltd.) by intravenous pump for 24 hours and 5 consecutive days.
  Interventions: Drug: Sivelestat sodium

INTERVENTIONS:
Drug: Sivelestat sodium — Continuous infusion of sivelestat sodium for 5 days
  Other Names: Mechanical ventilation

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by the host's maladjusted response to infection. It is one of the common clinical critical diseases, often accompanied by multiple organ failure, immune imbalance and high mortality. Sepsis is a syndrome of physiological, pathological and biochemical abnormalities caused by infection. Its incidence rate and prevalence have been on the rise in the past few years. Sepsis has greatly endangered the lives and health of the public. Among them, ARDS is a fatal complication of sepsis and a common critical illness syndrome in ICU. At present, the conventional treatment for ARDS caused by sepsis is still limited to indirect supportive therapy such as primary disease treatment, infection control, mechanical ventilation support, and nutrition improvement, lacking specific direct treatment methods. So far, the drug treatment effect of ARDS at home and abroad is not satisfactory. Therefore, it has become an urgent task to find a new treatment strategy to alleviate ARDS. Neutrophil elastase inhibitors can reversibly and competitively inhibit the release of neutrophil elastase, inhibit the activation of neutrophils and the infiltration of inflammatory cells in the lungs, alleviate the release of inflammatory mediators, and thus improve respiratory function, which has a good protective effect on various experimental ARDS. However, the efficacy of neutrophil elastase inhibitor represented by sivelestat sodium in the treatment of ARDS has reached a relatively consistent positive conclusion in animal experiments, while the results of clinical studies are different. These differences in clinical research still need further analysis, research and verification in clinical trials.

At present, the clinical studies of neutrophil elastase inhibitors in the treatment of sepsis induced ARDS are very few, and there is a lack of related prospective randomized controlled clinical studies. Therefore, further prospective clinical trials are needed to evaluate the therapeutic effect of neutrophil elastase inhibitors on sepsis induced ARDS patients. This study is intended to determine whether neutrophil elastase inhibitor can reduce the mechanical ventilation time, Murray lung injury score, ICU hospitalization time and 28-day mortality of septic ARDS patients compared with the control group through a single center randomized controlled trial, so as to provide a new basis for the treatment strategy of septic ARDS patients.

DETAILED DESCRIPTION:
Research content:

Randomized ARDS patients with mechanical ventilation caused by sepsis in the ICU were divided into test group (sivelestat sodium group) and control group (saline control group) according to 1:1 ratio. The mechanical ventilation time, lung injury score, ICU hospitalization time and 28-day mortality of the two groups were compared. Through statistical analysis, it was determined whether sivelestat sodium could reduce the mechanical ventilation time, lung injury score, ICU hospitalization time and 28-day mortality of ARDS patients caused by sepsis compared with the control group.

Research method and design scheme:

1. Study Design: Single center, randomized, blind, parallel controlled study.
2. Study population:

The patients with ARDS mechanical ventilation caused by sepsis admitted to the ICU of the First Hospital of Jilin University, aged 18-75 years, who can provide informed consent. According to sepsis 3.0, sepsis is a life-threatening organ dysfunction caused by the uncontrolled response of the body to infection. The diagnosis of ARDS is based on the Berlin definition.

(3) Intervention method:

1. Simple random grouping method (excel) is used to randomly assign patients who meet the inclusion criteria by 1:1. The specific method is: open excel, enter patient number (1-100) in the first column, enter "=RANDBETWEEN (1,2)" in the first case of the second column, and pull down to complete the inclusion code of all patients. 1 is the test group and 2 is the control group. According to the previous research results, based on the time of mechanical ventilation (days), the sample size was calculated using the mean comparison formula of two groups of independent samples. The mean value of the test group was 6.6, the standard deviation of the test group was 6.1, the mean value of the control group was 11.1, and the standard deviation of the control group was 8.4, α=0.05, β= 0.2. The sample size of the test group and the control group was calculated as 42 cases respectively. To prevent the sample from falling off, 100 cases were proposed to be included in the group, 50 cases in the test group (sivelestat sodium group) and 50 cases in the control group (saline control group).
2. Blinding method: after the intervention measures were implemented, the subjects were blinded, and sivelestat sodium and 0.9% sodium chloride were pumped intravenously in a uniform opaque packaging container.

(4) Administration method:

1. The patients in the test group were given 0.2 mg/kg. h of sivelestat sodium (0.1 g/tube, Shanghai Huilun Jiangsu Pharmaceutical Co., Ltd.) (the daily dose was added to 250 ml of 0.9% sodium chloride) intravenously for 24 hours and 5 consecutive days.
2. The patients in the control group were given 250 ml 0.9% sodium chloride (250ml/bag, Jilin Dubang Pharmaceutical Co., Ltd.) by intravenous pump for 24 hours and 5 consecutive days.

(5) Collect and observe indicators:

The demographic data (gender, age, height, weight), complications, APACHE II score, SOFA score, PCT, leukocytes, platelets, liver function, Murray lung injury score (Table 2), PaO2/FiO2, renal function, coagulation routine, Interleukin-2/4/6/10, mean arterial pressure, duration of mechanical ventilation, ICU hospitalization and 28-day survival were recorded.

(6) End point indicators:

1. Primary outcome: The duration of mechanical ventilation was compared between the two groups.
2. Secondary outcomes: Murray lung injury score, ICU hospitalization time and 28- day mortality were compared between the two groups.

(7) Statistical analysis:

SPSS 22.0 statistical software was used. The measurement data of normal distribution were expressed as mean ± standard deviation (x ± s), and the measurement data of non-normal distribution were expressed as median (interquartile interval). The pairwise comparison between groups was performed by t test or Mann Whitney U test; The chi square test or Fisher exact probability method was used to compare the counting data; To compare whether there is statistical difference in the end point indicators between the test group and the control group. Kaplan Meier survival curve was used to analyze and compare the difference of 28- day mortality between the two groups. P<0.05 was considered as the difference with statistical significance.

ELIGIBILITY:
Inclusion Criteria:

- 1. Adults (aged 18-75)

2. Patients with ARDS caused by sepsis

3. Patients admitted to ICU and mechanically ventilated

4. Patients who can provide informed consent

Exclusion Criteria:

* 1. Pregnant or lactating women;

  2. Patients allergic to planned medication;

  3. Patients who are expected to stay in the ICU for less than 5 days;

  4. Patients included in other trial items;

  5. Other reasons that the researcher thinks are not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation time | 2 years
  Comparison of mechanical ventilation time between the two groups

SECONDARY OUTCOMES:
Murray Lung Injury Score | 2 years
  Comparison of Murray lung injury scores between the two groups
ICU length of stay | 2 years
  Comparison of ICU length of stay between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Dong Zhang, doctor, Study Director — The First Hospital of Jilin University

IPD SHARING:
Plan to Share IPD: No
Not decided.

REFERENCES:
- [Result] Miyoshi S, Hamada H, Ito R, Katayama H, Irifune K, Suwaki T, Nakanishi N, Kanematsu T, Dote K, Aibiki M, Okura T, Higaki J. Usefulness of a selective neutrophil elastase inhibitor, sivelestat, in acute lung injury patients with sepsis. Drug Des Devel Ther. 2013 Apr 10;7:305-16. doi: 10.2147/DDDT.S42004. Print 2013. PMID 23596346
- See also: Usefulness of a selective neutrophil elastase inhibitor, sivelestat, in acute lung injury patients with sepsis — http://pubmed.ncbi.nlm.nih.gov/23596346/